CLINICAL TRIAL: NCT03833206
Title: A Phase I/II Study of PDC-1421 for Treating Depression in Cancer Patients: Part I Dose Escalation
Brief Title: A Phase I/II Study of PDC-1421 for Treating Depression in Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Collaborators: American BriVision Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABV-1601-001
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 PDC-1421 Capsule (Experimental): 1 PDC-1421 Capsule, trice daily, p.o. after meal for 28 days
  Interventions: Drug: PDC-1421 Capsule
- 2 PDC-1421 Capsules (Experimental): 2 PDC-1421 Capsule, trice daily, p.o. after meal for 28 days
  Interventions: Drug: PDC-1421 Capsule

INTERVENTIONS:
Drug: PDC-1421 Capsule — PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.

SUMMARY:
The purpose of this study is to evaluate the safety and the effective doses of PDC-1421 in cancer patients with depression.

ELIGIBILITY:
Eligibility Criteria

* 21 to 85 Years of age
* Diagnosis of Stage I, II or III cancer
* Histologically-proven malignancy
* Receiving or within one year of having received cancer treatment with radiation and/or chemotherapy
* Montgomery and Åsberg Depression Rating Scale (MADRS) ≥ 20 (moderate to severe depressive symptoms)
* Duration of depressive symptoms ≥ 2 weeks by patient report.
* No active/acute suicidality requiring immediate care or psychiatric hospitalization
* Sufficient English language proficiency to complete all assessments without assistance
* Able to swallow pills
* No severe anemia, defined as hemoglobin < 10 g/dL
* No history of multiple adverse drug reactions or allergy to study drugs
* Not pregnant
* No history of head trauma
* No history of epilepsy
* No other concurrent antidepressant medications

Exclusion Criteria

* Have a current or previous diagnosis of or history consistent with obsessive-compulsive disorder, posttraumatic stress disorder, bipolar I or II, manic or hypomanic episodes, schizophrenia, major Axis II disorders which might compromise the study, or major depression with psychotic symptoms, as assessed using the MINI International Neuropsychiatric Interview (MINI Plus).
* Have a documented history of an intellectual disability.
* Use of any antidepressant medication in the last 2 weeks before visit 1 (4 weeks for fluoxetine).
* Currently being treated with tamoxifen.
* Subjects who were non-responsive to two or more courses of antidepressant medications given at an adequate dosage* for symptom treatment within four weeks, or by the judgment of the investigator considered to have treatment resistant depression (TRD), or a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS) or psychosurgery within the last year.
* Have a history of any seizure disorder.
* Any clinically significant abnormal vital sign, ECG, or laboratory values as determined by the investigator which might interfere with the study.
* Have a high suicidal risk as assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS). High suicidal risk is indicated by:

  1. A positive response to question 4 or 5, indicating endorsement of suicidal ideation with at least some intent to act in the past month; and/or
  2. A positive response to part two of question 6, indicating the presence of any suicidal behavior in the past 3 months.
* Have a history of substance dependence/abuse** within the past 6 months or a positive drug screen result during the screening period.
* Have a history of severe allergies to more than 1 class of medication or multiple adverse drug reactions.
* * An adequate dosage of the antidepressant medication is defined as the average of the usual dose (mg/day) recommended in American Psychiatric Association (APA) Practice Guideline for the Treatment of Patients with Major Depressive Disorder, Third Edition. E.g. the usual dose of Citalopram is 20-60 mg/day, the adequate dosage is 40 mg/day.
* ** Tobacco is excluded here, and alcohol abuse is defined as average pure alcohol intake is more than 112 g (for male) or 56 g (for female) per week and/or with Alcohol withdrawal syndrome. Pure alcohol intake =% (Concentration or alcohol content) x c.c. (volume)x 0.79 (density of alcohol). Result of serum ethanol test should be equal to or lower than 10.0 mg/dL to be determined as eligible for the trial. If test result is between 10.1 to 29.9 mg/dL, only one re-test is allowed per subject to meet the criterion. Subject with test result equal to or higher than 30.0 mg/dL is to be excluded.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 5 weeks
  Change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline to week 1, 2, 3, 4, and 5 in patients taking 1 or 2 PDC-1421 capsules. The MADRS is a 10-item checklist including 1) depression [apparent]; 2) depression [reported]; 3) loss of interest; 4) suicidal ideation; 5) tension; 6) reduced appetite; 7) insomnia; 8) difficulty in activities; 9) concentration; and 10) pessimism. The MADRS is administered by a trained interviewer. Each item is rated on a scale of 0-6, with anchors at 2-point intervals; higher scores indicating more severity (i.e., ranging from 0 [no sadness] to 6 [extremely despondent]). The total score is used to define treatment response (≥50% reduction from baseline) and partial response (20-49% reduction from baseline). Remission is defined as a score of < 10. The following are used as an interpretation of scores:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression

CONTACTS AND LOCATIONS:
Overall Officials: scott A Irwin, MD/PhD, Principal Investigator — Cedars-Sinai Health System
Locations (1):
- Cedars-Sinai Health System, Los Angeles, California, United States